CLINICAL TRIAL: NCT03490578
Title: Effect of Robot-assisted Gait Training in Patients With Parkinson's Disease: a Randomized Controlled Trial
Brief Title: Robot-assisted Gait Training in Patients With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: National Rehabilitation Center, Seoul, Korea (Other Government)
Responsible Party: Principal Investigator, Han Gil Seo, Associate Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RAGT-PD1.0
Record Dates: First submitted 2018-03-21; First posted 2018-04-06 (Actual); Last update posted 2019-12-04 (Actual); Status verified 2019-12

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; Gait; Balance; Rehabilitation; Robot-assisted gait training
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robot-assisted gait training (Experimental): Robot-assisted gait training using an exoskeletal robot (Walkbot_S; P&S Mechanics Co. Ltd., Seoul, Korea)
  Interventions: Device: Robot-assisted gait training
- Intensive treadmill training (Active Comparator): Intensive treadmill training using an usual treadmill
  Interventions: Device: Intensive treadmill training

INTERVENTIONS:
Device: Robot-assisted gait training — Patients should use their belts (Harness) to support their weight when walking in equipment. In the first training session, the patient focuses on fitting and adapting the equipment and helps the patient learn. To minimize skin damage, the patient can wear a protector. The initial walking speed starts at 1.0 km/h and can be increased gradually to 3.0 km/h. The gait robot provides an auditory feedback according to gait cycle and a visual feedback on the patient's active participation. If the patient can tolerate, the gait robot may control the walking speed automatically according to the patient's participation. The treatment time per session is 45 minutes including don and doff time. Total 12 sessions are provided for 4 weeks.
  Arms: Robot-assisted gait training
Device: Intensive treadmill training — Patients exercise on the treadmill. The initial walking speed starts at 1.0 km/h and can be increased gradually to 3.0 km/h. The therapist provides appropriate visual and auditory instructions to allow the patient to participate in the treadmill training. The treatment time per session is 45 minutes including warm-up and cool-down. Total 12 sessions are provided for 4 weeks.
  Arms: Intensive treadmill training

SUMMARY:
Robot-assisted gait training can improve gait ability of patients with Parkinson's disease by repeating a normal gait pattern with high intensity. This study is a randomized controlled trial to investigate the effect of robot-assisted gait training on walking ability and functional connectivity of brain in patients with Parkinson's disease using an exo-skeletal robot.

DETAILED DESCRIPTION:
Parkinson's disease is a disease caused by dopamine deficiency in the striatum resulting from the loss of dopaminergic neuronal cells in the cerebral substantia. It is a progressive neurodegenerative disease characterized by motor symptoms including gait disturbance and balance instability. In the early stages of Parkinson's disease, dysfunction of the sensorimotor area of the basal ganglia typically occurs, leading to habitual control hurdles. Accordingly, cognitive efforts are required to perform habitual tasks such as walking, and the automaticity of walking is reduced. Walking performance in a dual-task condition has been used to assess gait automaticity in patients with Parkinson's disease.

Patients with Parkinson's disease are known to exhibit changes in functional connectivity of the brain from an early stage. In addition, a number of studies have reported that patients with Parkinson's disease with gait freezing have a change in resting brain activity and functional connectivity of the brain. However, no studies have examined the functional connectivity of the brain in patients with Parkinson's disease before and after rehabilitation.

Robot-assisted gait training is a method of rehabilitation that repeats normal gait patterns at high intensity. Recent meta-analysis has shown that robot-assisted gait training improved the recovery of independent gait after stroke compared with conventional rehabilitation therapy. On the other hand, robot-assisted gait training in Parkinson's disease has been reported to improve walking speed and walking endurance compared to conventional physical therapy, but is not superior to treadmill exercise of the same intensity. In addition, it has been reported that in patients with Parkinson's disease with balance impairment, robot-assisted gait training can improve balance disorder compared with physical therapy, and gait freezing has improved in some small-scale patients. However, studies on the effectiveness of robot-assisted gait training in Parkinson's disease are still lacking, and the mechanism of the effect has not been elucidated. In particular, the effect on gait automaticity, which is a characteristic of Parkinson 's disease, and functional connectivity of the brain has not been studied. Therefore, this study is aimed to investigate the effect of robot-assisted gait training on walking ability and functional connectivity of brain in patients with Parkinson's disease using an exo-skeletal robot.

ELIGIBILITY:
Inclusion Criteria:

* Clinically confirmed patients with idiopathic Parkinson's disease
* Hoehn & Yahr stage 2.5 or 3 patients
* Patients with a Mini-Mental Status Examination (MMSE) score of 24 or higher

Exclusion Criteria:

* Patients with severe dyskinesia or on-off fluctuations due to medication
* Patients who need to change drugs during the study period
* Patients with sensory abnormalities of the lower limb
* Patients with vestibular disease or paroxismal vertigo
* Patients with other neurological or orthopedic disease involving legs, or severe cardiovascular diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2018-04-23 (Actual); Primary Completion 2019-11-14 (Actual); Study Completion 2019-11-14 (Actual)

PRIMARY OUTCOMES:
10 meter walk test (sec) : single task | at 4 weeks

SECONDARY OUTCOMES:
10 meter walk test (sec) : single task | baseline, at 8 weeks
10 meter walk test (sec) : cognitive dual-task | baseline, at 4 weeks, at 8 weeks
10 meter walk test (sec) : physical dual-task | baseline, at 4 weeks, at 8 weeks
Berg balance scale | baseline, at 4 weeks, at 8 weeks
  The Berg balance scale is used to objectively determine a patient's ability (or inability) to safely balance during a series of predetermined tasks. It is a 14 item list with each item consisting of a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of function (Maximum score 56).
Timed-up & go test (sec) | baseline, at 4 weeks, at 8 weeks
Korean version of Falls Efficacy Scale-International | baseline, at 4 weeks, at 8 weeks
  The FES-I is a 16-item questionnaire of fall-related self-efficacy. The 16 items of the FES-I are rated according to "how concerned you are about the possibility of falling", using the following responses (score in parentheses): not at all (1), somewhat (2), fairly (3), and very concerned (4). Thus, the total score ranges from 16 to 64 points.
New Freezing of Gait questionnaire (NFOG-Q) - Part I | baseline, at 4 weeks, at 8 weeks
  Part I detected the presence of FOG using a dichotomous item in which individuals were classified as a freezer (FR) or a non-freezer (NFR) if they had experienced FOG-episodes during the past month.
New Freezing of Gait questionnaire (NFOG-Q) - Part II, III | baseline, at 4 weeks, at 8 weeks
  Parts II and III were designed for FRs only, providing a total summed score between 0 and 28. Part II (items 2-6, scoring range 0-19) rated the severity of FOG based on its duration and frequency in its most common manifestation, i.e. during turning and initiation of gait. Part III rated the impact of FOG on daily life (items 7-9, scoring range 0-9). No separate on and off rating of parts II and III was considered to avoid unreliable assessment.
Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPRDS) - Part I | baseline, at 4 weeks, at 8 weeks
  Part I - Non-motor experiences of daily living, questionnaire
Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPRDS) - Part II | baseline, at 4 weeks, at 8 weeks
  Part II - Motor experiences of daily living, questionnaire
Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPRDS) - Part III | baseline, at 4 weeks, at 8 weeks
  Part III - Motor examination, structured physical examination
Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPRDS) - Part IV | baseline, at 4 weeks, at 8 weeks
  Part IV - Motor complications, questionnaire
Functional connectivity in resting-state fMRI (Correlation coefficient) | baseline, at 4 weeks
  * Correlation coefficient between BOLD signals in motor network
  * At least 6 minutes resting state fMRI imaging is desirable for acquiring stable resting state brain imaging data. The investigators divide the entire brain into voxels, and if the investigators assume TR=3sec, one voxel has 120 time series data. This data reflects the blood-oxygenation level dependent (BOLD) signal, which is related to neural activity via a complex interplay of cerebral blood flow, blood volume, and metabolic rate of oxygen.

CONTACTS AND LOCATIONS:
Overall Officials: Han Gil Seo, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Kim H, Kim E, Yun SJ, Kang MG, Shin HI, Oh BM, Seo HG. Robot-assisted gait training with auditory and visual cues in Parkinson's disease: A randomized controlled trial. Ann Phys Rehabil Med. 2022 May;65(3):101620. doi: 10.1016/j.rehab.2021.101620. Epub 2022 Feb 23. PMID 34896605
- [Derived] Kang MG, Yun SJ, Shin HI, Kim E, Lee HH, Oh BM, Seo HG. Effects of robot-assisted gait training in patients with Parkinson's disease: study protocol for a randomized controlled trial. Trials. 2019 Jan 7;20(1):15. doi: 10.1186/s13063-018-3123-4. PMID 30616685